CLINICAL TRIAL: NCT03333395
Title: Efficacy of Nebulized Heparin and Salbutamol in Mechanically Ventilated Patients With Acute Exacerbation Chronic Obstructive Pulmonary Disease: a Randomized Clinical Trial
Brief Title: Nebulized Heparin and Salbutamol in Mechanically Ventilated Patients With AECOPD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Dr.Ibrahim Mamdouh Esmat, Lecturer of Anesthesia and Intensive Care Department, Faculty of Medicine, Ain- shams University, Cairo, Egypt., Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R 26 / 2017
Record Dates: First submitted 2017-11-02; First posted 2017-11-06 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Mechanically Ventilated Patients
Keywords: Mechanical ventilation; Acute Exacerbation of chronic obstructive airway disease (AECOPD); Nebulized heparin; C-Reactive Protein (CRP
MeSH Terms: interventions — Albuterol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HS Group (study group) (Active Comparator)
  Interventions: Drug: Nebulized heparin and salbutamol
- S Group (control group) (Active Comparator)
  Interventions: Drug: Nebulized salbutamol

INTERVENTIONS:
Drug: Nebulized heparin and salbutamol — HS Group medications (study group) (30 patients) which was prepared by adding Heparin 25000 IU in 5ml (5 ampoules of Heparin Sodium 5000 I.U/ML, Nile company for Pharmaceuticals and Chemical Industries-A.R.E.) to Salbutamol 5mg/2.5ml Nebulizer Solution (one Ventolin nebule containing a preservative-free solution of Salbutamol Sulphate BP 2.5mg, GlaxoSmithKline Inc.)
  Arms: HS Group (study group)
Drug: Nebulized salbutamol — S Group medications (control group) (30 patients) which was prepared by adding Salbutamol 5mg/2.5ml Nebulizer Solution + Na cl 0.9% 5ml.
  Arms: S Group (control group)

SUMMARY:
This randomised study was designed to assess the efficacy of nebulised heparin and salbutamol in improving lung function in mechanically ventilated patients with AECOPD.

DETAILED DESCRIPTION:
Methods:

Patients:

This study was performed between February 2017 and September 2017. Admitted Patients to the Internal Medicine ICU of Ain-Shams University Hospitals were screened for meeting enrollment criteria. Written informed consent was taken from all patients, their parents or their guardians before any study procedure was done. Patients were included in the study if they were > or = 18 years of age, body weight 70-110Kg, height 160-180 cm with clinically evident AECOPD and in need for mechanical ventilation confirmed by arterial blood gases (ABGs).

Excluded Patients from the study were those who were not enrolled within the first 24 hours of mechanical ventilation and those who were likely to be extubated within 24 hours. Patients were also excluded if they have any history of ischemic heart disease, pulmonary bleeding within the previous 3 months, history of bleeding diathesis, known to be allergic to heparin or history of thrombocytopenia after previous treatment with heparin. Female patients were excluded if they are pregnant or breast feeding.

Study design:

This study was a double-blind, randomized controlled trial. Block randomization was performed in random blocks of two to eight. After enrollment, patients were randomly allocated into either of the two groups, HS and S. Allocations were concealed in opaque, sequentially numbered, sealed envelopes.

Study medications:

Patients in either group were treated by nebulization of 7.5 ml of study medication every 6 hours (4imes a day). The study medications were prepared by the local pharmacist who gave them to the nurse in charge and they were not involved in any other part of the study.

The study medications were either a HS Group medications (study group) (30 patients) which was prepared by adding Heparin 25000 IU in 5ml (5 ampoules of Heparin Sodium 5000 I.U/ML, Nile company for Pharmaceuticals and Chemical Industries-A.R.E.) to Salbutamol 5mg/2.5ml Nebulizer Solution (one Ventolin nebule containing a preservative-free solution of Salbutamol Sulphate BP 2.5mg, GlaxoSmithKline Inc.) or S Group medications (control group) (30 patients) which was prepared by adding Salbutamol 5mg/2.5ml Nebulizer Solution + Na cl 0.9% 5ml.

Standard medications were used in both groups which included analgesics, sedatives, fluid management, antibiotic prophylaxis, steroids and thrombo-prophylaxis according to local guidelines.

Nebulization and Ventilation:

Nebulization was conducted by adding the nebulization medication to a nebulization chamber (Ameco Technology, particle size 0.5 To 10um, Nebulization rate> 0.3ml/min) connected to the inspiratory limb of the breathing circuit by a T-piece (22M-22M/15F, with port- TNTAIR medical) close to the patient but after the moist exchanger if applied. An expiratory filter was applied in the expiratory limb of the breathing circuit. The nebulization session was continued for at least 20 minutes.

Patients in the heparin group were eliminated (drop-out) if they developed a heparin-induced thrombocytopenia, an increase in APTT more than double normal,an evident bleeding that necessitated blood transfusion or if an excessive blood tinged sputum or bleeding appeared during suctioning or bronchial lavage.

All patients were mechanically ventilated using SIMV mode, with a targeted TV: 6-8 ml/kg, rate: 10-12 bpm, PEEP: 5-10 cm H2O, and FIO2:40%-60%.

Data collection:

The PaO2/FiO2 ratio and, PaCo2 were measured each day at 7 a.m. No changes in the ventilator settings or the patient's position were permitted for the 10 minutes before this measurement.

Demographic data including history of smoking (never, former, current) were collected on study entry, and ventilation parameters, clinical and radiological data, sputum character, medication usage, and adverse events, including blood-stained sputum or frank blood in sputum and red cell transfusions, were recorded daily while the patient remained mechanically ventilated.

Ventilator- free days were defined as the number of days patients were breathing without mechanical ventilation during the first 14 days.

Development of acute lung injury (ALI) was defined using the consensus criteria (15). Vasopressor usage was defined by the administration of any of the following: dopamine, dobutamine, norepinephrine, or epinephrine. Renal failure was defined as a serum creatinine of greater than 300 μmol/L or urine output of less than 500 mL per day or renal replacement therapy for acute renal impairment. Respiratory failure was defined as the acute requirement for mechanical ventilation primarily due to acute exacerbation of COPD evident clinically by severe shortness of breath, with or without Co2 narcosis, and by ABG as PH <7.3, PaO2<60 mmHg and PaCO2 >50 mmHg.

Outcomes:

The following data were collected and compared for each group with respect to:

The primary outcome was:

* The number of ventilator hours; number of hours during which the patient was mechanically ventilated.
* The average daily ratio of partial pressure of oxygen to FiO2 (PaO2/FiO2) while the patient remained ventilated for a maximum of 14 days from randomization and

The secondary outcome was:

* The length of ICU stays.
* CRP quantitative titer was measured daily as part of the routine clinical care. The maximum serum CRP level during the ICU stay was designated as max- CRP as a prognostic factor. Normal concentration of CRP in healthy human serum is between 5 and 10 mg/L, increasing with aging(14).
* Platelets count and
* The number of suctions with blood tinged sputum.

Analysis of Data:

Depending on Dixon et al.,2010(16) who found that the ventilation free days (22.6 ±4.0 and 18.0 ± 7.1 in heparin and control groups respectively, and assuming the power= 0.80 and α=0.05, and by using PASS 11th release the minimal sample size for an equal size controlled clinical trial is 26 in each group. We will recruit 30 in each group for possible attrition (17,18).

The collected data were coded, tabulated, and statistically analyzed using IBM SPSS statistics (Statistical Package for Social Sciences) software version 22.0, IBM Corp., Chicago, USA, 2013.

ELIGIBILITY:
Inclusion Criteria:

* > or = 18 years of age,
* body weight 70-110Kg,
* height 160-180 cm
* with clinically evident AECOPD and in need for mechanical ventilation confirmed by arterial blood gases (ABGs).

Exclusion Criteria:

* Excluded Patients from the study were those who were not enrolled within the first 24 hours of mechanical ventilation and those who were likely to be extubated within 24 hours. - History of ischemic heart disease,
* History of pulmonary bleeding within the previous 3 months,
* History of bleeding diathesis,
* Known to be allergic to heparin or
* History of thrombocytopenia after previous treatment with heparin.
* Female patients were excluded if they were pregnant or breast feeding.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
The number of ventilator hours | Maximum of 14 days from randomization.
  Number of hours during which the patient was mechanically ventilated.

CONTACTS AND LOCATIONS:
Locations (1):
- Internal Medicine ICU of Ain-Shams University Hospitals, Cairo, Egypt